CLINICAL TRIAL: NCT03429049
Title: A Randomized, Double-blind, Placebo-controlled, Single Injection, 52-Week Study to Evaluate the Efficacy and Safety of an Intra-articular Injection of CNTX-4975-05 in Subjects With Chronic, Moderate-to-severe Osteoarthritis Knee Pain
Brief Title: A Phase 3 Efficacy and Safety Study of Intra-articular CNTX-4975-05 (Capsaicin) vs Placebo in Subjects With OA Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNTX-4975i-OA-301
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
Keywords: analgesic; non-opioid; capsaicin; intra-articular; osteoarthritis; pain; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo of 2.0 mL for IA injection
  Interventions: Drug: Placebo
- CNTX-4975-05 (Experimental): Pre-filled glass syringes administered as a single 2.0 mL IA injection
  Interventions: Drug: CNTX-4975-05

INTERVENTIONS:
Drug: CNTX-4975-05 — Receiving CNTX-4975-05 injection
  Arms: CNTX-4975-05
Drug: Placebo — Receiving Placebo injection
  Arms: Placebo

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled, single injection, 52-week study to evaluate the analgesic efficacy and safety of a single intra-articular (IA) CNTX-4975-05 (capsaicin), compared to IA placebo, in subjects with chronic, moderate-to-severe osteoarthritis (OA) knee pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects between 40 and 95 years of age (inclusive) at the time of the Screening Visit with the ability to comply with answering the electronic diary using the study-provided tablet computers.
* Confirmation of osteoarthritis (OA) of the knee.
* Confirmation of OA of the index knee.
* Moderate to severe pain in the index knee associated with OA must be stable for a minimum of 6 months prior to Screening, as assessed by the investigator.
* BMI ≤45 kg/m^2.
* Must have failed 2 or more prior therapies.
* Females not of childbearing potential, defined as post-menopausal for at least 1 year, or surgically sterile, or practicing one of the following medically acceptable methods of birth control throughout the study period.
* Subject agrees to stay on their current pain medication (including over the counter (OTC) medications) from the time of Screening through Week 12. The current pain medication must be taken only for pain in the index knee, and not for another pain indication.
* Subject agrees to take only the allowed rescue medications for OA knee pain of the index knee from the time of Screening through study completion and agrees to use no topical medications for OA knee pain during the trial.

Key Exclusion Criteria:

* Joint replacement surgery of the index knee at any time, or open surgery of the index knee in the past 24 months.
* Prior arthroscopic surgery of the index knee within 6 months of Screening.
* Any painful conditions of the index knee due to joint disease other than OA.
* Periarticular pain from any cause.
* Pain in the non-index knee that is >3 on a numeric pain rating scale (NPRS) (0-10) when walking or at rest.
* Other chronic pain anywhere in the body that requires the use of analgesic medications.
* Instability of the index knee.
* Misalignment (>10 degrees varus or valgus) of the index knee on standing.
* Documented history of neuropathic arthropathy or finding of bony fragmentation in the index knee with imaging.
* Physical/ occupational/ chiropractic therapy for the lower extremities or acupuncture for the lower extremities within 30 days of Screening, or need for such therapy during the study.
* Plans to have surgery, other invasive procedures, or IA injections while participating in the study.
* Has used topical capsaicin on the index knee within 90 days of Screening.
* Current use of opioids for any condition other than for OA of the index knee.
* Corticosteroid injection into the index knee within 90 days of Screening.
* Received IA viscosupplementation (eg, Synvisc®, Hyalgan®) within 90 days of Screening.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall M. Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (33):
- United States (33):
  - Alabama Orthopaedic Center - Research, Birmingham, Alabama
  - Cahaba Research, Inc, Birmingham, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Noble Clinical Research, LLC, Tucson, Arizona
  - Orange County Research Institute, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Providence Clinical Research, North Hollywood, California
  - Medical Associates Research Group, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Tampa Bay Medical Research, Inc, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - M&M Medical Center, Inc, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Jewett Orthopaedic, Orlando, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Atlanta Orthopaedic Institute, LLC, Stockbridge, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Mid America PolyClinic, Overland Park, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Tristan Medical Enterprises PC, dba, North Attleboro, Massachusetts
  - Medical Research Associates, Inc, Traverse City, Michigan
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bone Joint & Spine Surgeons, Inc, Toledo, Ohio
  - Tekton Research, Inc, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Ortho Virginia, Arlington, Virginia
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | CNTX-4975-05
Started | 138 | 194
Treated | 136 | 189
Completed | 110 | 152
Not Completed | 28 | 42
Not completed — Adverse Event | 2 | 3
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 4 | 2
Not completed — Lost to Follow-up | 9 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Sponsor Decision | 2 | 0
Not completed — Withdrawal by Subject | 4 | 20
Not completed — Other reasons: UNABLE TO ADMINISTER IP, COLLECT ASPIRATE | 3 | 8

BASELINE CHARACTERISTICS:
Population: The safety population is defined as any subject that received any amount of investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CNTX-4975-05 | Total
Number analyzed (Participants) | 136 | 189 | 325
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (9.5) | 61.8 (9.1) | 61.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 123 | 206
  Male | 53 | 66 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 37 | 60
  Not Hispanic or Latino | 113 | 152 | 265
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 15 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 46 | 76
  White | 90 | 123 | 213
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 4 | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.07 (5.801) | 31.55 (5.692) | 31.77 (5.734)
Baseline Pain with Walking NPRS (0-10) Score [Mean (Standard Deviation); unit: score on a scale] — Average daily OA pain in the index knee while walking was evaluated using a 0 to 10 Numerical Pain Rating Scale (NPRS) (0 = no pain and 10 = worst possible pain). 0 was the best score and 10 was the worst score.
  score on a scale | 7.09 (1.152) | 7.06 (1.082) | 7.07 (1.110)
Baseline WOMAC A (Pain) Domain Score (range 0-50) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The pain dimension includes 5 items about the amount of pain experienced doing various activities (walking, stair climbing, nocturnal, at rest, weight bearing). The score ranges from 0 to 50. 0 being the best score and 50 being the worst.
  score on a scale | 30.80 (8.166) | 31.92 (7.493) | 31.45 (7.788)
Baseline WOMAC B (Stiffness) Domain Score (range 0-20) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The stiffness dimension includes 2 items about the joint stiffness upon wakening and joint stiffness later in the day. The score ranges from 0 to 20. 0 being the best score and 20 being the worst.
  score on a scale | 13.24 (3.389) | 13.28 (3.232) | 13.26 (3.293)
Baseline WOMAC C (Function) Domain Score (range 0-170) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The physical function dimension asks about the degree of difficulty in doing 17 activities due to the reference joint. The score ranges from 0 to 170. 0 being the best score and 170 being the worst.
  score on a scale | 105.25 (29.755) | 108.23 (27.085) | 106.99 (28.222)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Weekly Pain With Walking (NPRS 0-10) in the Index Knee
Description: Average daily OA pain in the index knee while walking was evaluated using a 0 to 10 Numerical Pain Rating Scale (NPRS) (0 = no pain and 10 = worst possible pain). 0 was the best score and 10 was the worst score.
  Subjects used an ePRO at bedtime (9:00 PM ± 3 hours) to record on a daily basis their average daily OA knee pain score with walking during the previous 24 hours.
Time Frame: Baseline, Week 12
Population: The intent to treat (ITT) population included all randomized subjects who received any amount of investigational product and all observed data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 130 | 177
score on a scale | -2.84 (0.212) | -3.17 (0.182)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; The NRS least squares mean difference in change from baseline between treatment arms was analyzed with a mixed model for repeated measures (MMRM). It included terms for treatment, pooled study center, baseline K L grade category for the index knee, baseline BMI category, sex, study week, treatment by visit study week interaction, and baseline average daily pain with walking NPRS (0-10) score as covariates, using an unstructured covariance structure; Test type: Superiority; p = 0.1904, Mixed Models Analysis; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.84 to 0.17], Standard Error of Mean 0.256

2. Secondary Outcome: Mean Change From Baseline in WOMAC A (Pain) Dimension Total Score
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The pain dimension includes 5 items about the amount of pain experienced doing various activities (walking, stair climbing, nocturnal, at rest, weight bearing). The score ranges from 0 to 50.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 128 | 174
score on a scale | -12.72 (1.002) | -15.42 (0.860)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; The WOMAC A least squares mean difference in change from baseline between treatment arms was analyzed with a mixed model for repeated measures (MMRM). It included terms for treatment, pooled study center, baseline K L grade category for the index knee, baseline BMI category, sex, study week, treatment by visit study week interaction, and baseline average daily pain with walking NPRS (0-10) score as covariates, using an unstructured covariance structure; Test type: Superiority; p = 0.0257, Mixed Models Analysis; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-5.07 to -0.33], Standard Error of Mean 1.206

3. Secondary Outcome: Mean Change From Baseline WOMAC B (Stiffness) Dimension Total Score
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The stiffness dimension has 2 items: joint stiffness upon wakening and joint stiffness later in the day. The score ranges from 0 to 20.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 128 | 174
score on a scale | -5.21 (0.448) | -6.15 (0.386)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; The WOMAC B least squares mean difference in change from baseline between treatment arms was analyzed with a mixed model for repeated measures (MMRM). It included terms for treatment, pooled study center, baseline K L grade category for the index knee, baseline BMI category, sex, study week, treatment by visit study week interaction, and baseline average daily pain with walking NPRS (0-10) score as covariates, using an unstructured covariance structure; Test type: Superiority; p = 0.0855, Mixed Models Analysis; Least Squares Mean Difference = -0.94, 95% CI 2-sided [-2.01 to 0.13], Standard Error of Mean 0.545

4. Secondary Outcome: Mean Change From Baseline in WOMAC C (Physical Function) Dimension Total Score
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The function dimension asks about the degree of difficulty in doing 17 activities due to the reference joint. The score ranges from 0 to 170.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 128 | 174
score on a scale | -42.70 (3.417) | -50.49 (2.935)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; The WOMAC C least squares mean difference in change from baseline between treatment arms was analyzed with a mixed model for repeated measures (MMRM). It included terms for treatment, pooled study center, baseline K L grade category for the index knee, baseline BMI category, sex, study week, treatment by visit study week interaction, and baseline average daily pain with walking NPRS (0-10) score as covariates, using an unstructured covariance structure; Test type: Superiority; p = 0.0550, Mixed Models Analysis; Mean Difference (Final Values) = -7.80, 95% CI 2-sided [-15.86 to 0.26], Standard Error of Mean 4.096

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Placebo | CNTX-4975-05
All-Cause Mortality (participants affected / at risk) | 0/136 | 1/189
Serious Adverse Events (participants affected / at risk) | 6/136 | 6/189
Other Adverse Events (participants affected / at risk) | 45/136 | 110/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=136) | CNTX-4975-05 (N=189)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response (General disorders) | 0 (0) | 1 (1)
Oestrogen receipt positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Branchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=136) | CNTX-4975-05 (N=189)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 19 (19)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 8 (8)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4)
Influenza (Infections and infestations) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 12 (12)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Injection site joint pain (General disorders) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03429049/Prot_SAP_000.pdf